CLINICAL TRIAL: NCT00024193
Title: A Study Of The Treatment Of Metastatic Neuroblastoma In Children More Than One Year Of Age At Diagnosis
Brief Title: Chemotherapy and Surgery Followed by Peripheral Stem Cell Transplantation in Treating Patients With Metastatic Neuroblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Collaborators: Societe Francaise Oncologie Pediatrique (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CCLG-NB-1999-02; CDR0000068899 (Registry Identifier: PDQ (Physician Data Query)); SFOP-NB97; EU-20106
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2001-11

CONDITIONS: Neuroblastoma
Keywords: stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Busulfan; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Melphalan; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: melphalan
Drug: vincristine sulfate
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs to kill more tumor cells. Chemotherapy, given before and after surgery, followed by peripheral stem cell transplantation may be an effective treatment for metastatic neuroblastoma.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy, given before and after surgery, followed by peripheral stem cell transplantation in treating patients who have metastatic neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of induction chemotherapy followed by surgical resection and consolidation chemotherapy with autologous peripheral blood stem cell transplantation in patients with metastatic neuroblastoma.
* Determine the tolerability and feasibility of this regimen in these patients.
* Determine the medium and long-term results in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive induction chemotherapy comprising cyclophosphamide IV over 6 hours on days 1 and 2 and doxorubicin IV continuously and vincristine IV continuously over days 1-3 of courses 1, 2, 4, and 6. Patients receive cisplatin IV over 1 hour on days 1-4 and etoposide IV over 2 hours on days 1-3 of induction courses 3, 5, and 7. Patients also receive filgrastim (G-CSF) IV or subcutaneously once daily beginning on day 5 of courses 3, 5, and 7 and continuing until blood counts recover. Treatment repeats every 21 days.

At the completion of induction chemotherapy, patients undergo surgical resection. Patients in complete remission receive high-dose consolidation chemotherapy comprising oral busulfan every 6 hours on days -7 to -3 and melphalan IV over 2 minutes on day -2. Autologous peripheral blood stem cells (PBSC) are reinfused on day 0. Patients with n-myc tumor amplification undergo radiotherapy at least 70 days after PBSC transplantation.

Patients are followed every 6 months.

PROJECTED ACCRUAL: Approximately 15-45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed primary neuroblastoma OR
* Presence of neuroblasts in bone marrow associated with an elevation of urinary catecholamines
* Metastatic disease demonstrated by at least 1 of the following:

  * Medullary invasion (bone marrow involvement) as indicated by bone uptake on meta-iodobenzyl guanidine I 123 or bone lesions on bone scan
  * Distant metastases to liver, pleura, lungs, or distant nodes
* No 11-22 translocation

PATIENT CHARACTERISTICS:

Age:

* 1 and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* See Disease Characteristics

Other:

* No contraindications to study drugs

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-04

CONTACTS AND LOCATIONS:
Overall Officials: Janice A. Kohler, MD, FRCP, Study Chair — University Hospital Southampton NHS Foundation Trust; D. Valteau-Couanet, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Institut Gustave Roussy, Villejuif, France